CLINICAL TRIAL: NCT04725630
Title: A Healthy Food Prescription Incentive Program for Adults With Type 2 Diabetes Who Are Experiencing Food Insecurity
Brief Title: Healthy Food Prescription Incentive Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Alberta Health services (Other); Alberta Blue Cross (Unknown); Nu Skin Enterprises (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dana Lee Olstad, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB20-0543
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Diet, Healthy; Diabetes Mellitus, Type 2; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators will be blinded to group allocation during data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subsidized Healthy Food Prescription Incentive (Experimental): Participants will receive a one-time healthy food prescription pamphlet from their healthcare provider and a weekly incentive of $10.50/household member to purchase healthy foods in supermarkets for 12 months. The list of incentive-eligible foods includes whole, minimally processed foods with little to no added fat, sugar or salt from all food groups.
  Interventions: Behavioral: Healthy food incentive; Behavioral: Healthy food prescription
- Healthy Food Prescription Comparison (Active Comparator): Participants will receive a one-time healthy food prescription pamphlet from their healthcare provider. The pamphlet closely mimics current standard of care for patients with diabetes in Alberta (i.e., nutrition counselling).
  Interventions: Behavioral: Healthy food prescription

INTERVENTIONS:
Behavioral: Healthy food incentive — $10.50/week/household member for 12 months to purchase healthy foods in participating supermarkets.
  Arms: Subsidized Healthy Food Prescription Incentive
Behavioral: Healthy food prescription — A one-time healthy food prescription pamphlet

SUMMARY:
It is important for individuals with type 2 diabetes (T2DM) to adhere to a healthy dietary pattern to maintain optimal blood glucose levels and overall health. The increasing costs of healthy foods, however, is a barrier to maintaining healthful dietary patterns, particularly for individuals with T2DM who are experiencing food insecurity (i.e., inadequate or insecure access to food due to financial constraints). Lower diet quality may result in difficulties maintaining optimal blood glucose levels, leading to higher rates of diabetes complications, and increased acute care usage and costs.

Effective strategies to address this issue are lacking despite the well-known impact of food insecurity on maintaining optimal blood glucose levels. One way to address this problem is to provide incentives to purchase healthy foods through healthy food prescription programs. These programs may help to reduce food insecurity and improve diet quality, thereby improving blood glucose control and reducing diabetes complications over time.

This study will investigate the reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) of a healthy food prescription incentive program among adults who are experiencing food insecurity and persistent hyperglycemia through three concurrent studies; a randomized controlled trial, an implementation study, and a modelling study.

The randomized controlled trial will examine the effectiveness of a healthy food prescription incentive program compared to a healthy food prescription alone in reducing blood glucose levels among adults who are experiencing food insecurity and persistent hyperglycemia.

DETAILED DESCRIPTION:
It is vital for individuals with type 2 diabetes (T2DM) to adhere to a healthy dietary pattern to maintain optimal blood glucose levels and overall health. However, the increasing costs of healthy foods is a barrier to maintaining healthful dietary patterns, particularly for individuals with T2DM who are experiencing food insecurity (i.e., inadequate or insecure access to food due to financial constraints). Lower diet quality may result in difficulties maintaining optimal blood glucose levels, leading to higher rates of diabetes complications, and increased acute care usage and costs.

Although the adverse impact of food insecurity on maintaining optimal blood glucose levels is well documented, effective strategies to address food insecurity among individuals with T2DM are lacking. One approach to address this problem is to provide incentives for individuals to purchase healthy foods through healthy food prescription programs. These programs may help to reduce food insecurity and improve diet quality, thereby improving blood glucose levels and reducing diabetes complications over time.

Using a type 2 hybrid effectiveness-implementation design, we will conduct three concurrent studies (i.e. randomized controlled trial, implementation study, modelling study) to examine the reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) of a healthy food prescription incentive program among adults who are experiencing food insecurity and persistent hyperglycemia. The randomized controlled trial will examine the effectiveness of a healthy food prescription incentive program compared to a healthy food prescription alone in improving blood glucose levels, quantified via hemoglobin A1C, among adults who are experiencing food insecurity and persistent hyperglycemia. Secondary outcomes include blood glucose levels quantified via fructosamine, the proportion of patients with elevated hemoglobin A1C (i.e. ≥ 8.5%), diet quality and skin carotenoid levels, intermediate clinical outcomes (blood lipids, blood pressure, BMI, waist circumference, need for anti-hyperglycemic medication/insulin) and patient-reported outcomes (psychosocial well-being, self-rated health, diabetes self-efficacy, diabetes self-management, diabetes distress, diabetes competing demands, perceived financial barriers to chronic disease care, hypoglycemic episodes, household food insecurity).

Methods: 594 adults who are experiencing food insecurity and persistent hyperglycemia (i.e., hemoglobin A1C 6.5-12%) from urban and rural primary care clinics will be randomized to a 12 month healthy food prescription incentive (n=297) or a healthy food prescription comparison group (n=297).

The healthy food prescription incentive program consists of the following two core elements: 1) The one-time healthy food prescription pamphlet is a low literacy resource comprised of a pre-printed healthy food prescription that outlines an evidence-based healthy dietary pattern; 2) The healthy food incentive provides a weekly incentive of $10.50/household member to purchase healthy foods in participating supermarkets for 12 months. The intervention will be delivered over 12 months to allow sufficient time for dietary changes to be reflected in several A1c cycles.

At baseline (0 months) and follow-up (12 months), participants will access a pilot-tested web-based platform to provide responses to sociodemographic and health-related items, and a variety of patient-reported outcomes, including household food insecurity. To assess diet quality, dietary intake will be assessed via two 24-hour dietary recalls at each time point using the Automated Self-Administered Dietary Assessment Tool for Canada (ASA24-Canada-2018). Clinical measurements (biochemical and physical measurements) will be obtained to assess blood glucose, blood lipids, BMI, blood pressure, skin carotenoids, and waist circumference. Need for anti-hyperglycemic medication/insulin will be quantified via administrative health records. At 6 months and 18 months participants will have their blood glucose levels measured. They will also report their dietary intake via two 24-hour dietary recalls and their household food insecurity status.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-85 years) with type 2 diabetes (or diabetes of unknown etiology)
* Persistent hyperglycemia (i.e. hemoglobin A1C 6.5-12%)
* Are currently experiencing food insecurity and/or report that it is difficult/very difficult to make ends meet
* Can communicate in English or have someone to translate

Exclusion Criteria:

* A1c <6.5% or > 12% given the recommendation for anti-hyperglycemic treatment escalation for those with A1c>12%
* Reside in a facility that provides meals (e.g., shelter, long-term care, prison)
* Exhibit signs/symptoms of metabolic decompensation (weight loss, polyuria, polydipsia)
* Diagnosis of eating disorder(s) (e.g., anorexia nervosa, bulimia)
* Have experienced diabetic ketoacidosis or a hyperglycemic hyperosmolar emergency in the past year
* Experienced a hypoglycemic event in the past 3 months
* Are trying to conceive, pregnant and/or breastfeeding
* Are currently participating in other clinical trials
* A household member is currently or has previously participated in this trial
* Unwilling/unable to shop in study-affiliated supermarkets for the next 12 months
* Plan to leave for Canada for more than 2 weeks in the next 12 months
* Unable to complete data collection at follow-up (e.g., due to moving)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels via hemoglobin A1C | Assessed at Baseline (0 months) and Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in blood glucose levels measured by hemoglobin A1C

SECONDARY OUTCOMES:
Blood glucose levels via elevated hemoglobin A1C | Assessed at Baseline (0 months) and Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in proportion of patients with elevated hemoglobin A1C (>/=8.5%)
Blood glucose levels via fructosamine | Assessed at Baseline (0 months) and Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in blood glucose levels via fructosamine
Overall diet quality by Healthy Eating Index-2015 and by Healthy Eating Food Index-2019 | Assessed twice at Baseline (0 months) and twice at Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in mean diet quality by Healthy Eating Index-2015 scores and by Healthy Eating Food Index-2019 scores
Diet quality sub-scores by Healthy Eating Index-2015 and by Healthy Eating Food Index-2019 | Assessed twice at Baseline (0 months) and twice at Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in diet quality component scores by Healthy Eating Index-2015 and by Healthy Eating Food Index-2019
Fruit and vegetable intake via skin carotenoids | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in skin carotenoids
Blood Lipids | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in blood lipids including total-, HDL- and LDL-cholesterol, triglycerides, apolipoprotein B
Blood Pressure | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in both systolic and diastolic blood pressure
Body Mass Index | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in Body Mass Index
Waist Circumference | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in waist circumference
Anti-hyperglycemic Medication/Insulin | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in need for anti-hyperglycemic medication and/or insulin.
World Health Organization-5 Well-Being Scale scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in World Health Organization Well-Being Scale scores. The World Health Organization Well-Being scale will be used to assess experiences of well-being in the last 2 weeks with scores ranging from 0 (worst possible quality of life) to 25 (best imaginable quality of life).
Stanford Diabetes Self-efficacy Scale scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in Stanford Diabetes Self-efficacy Scale scores. The Stanford Diabetes Self-efficacy Scale will be used to assess confidence in completing activities related to diabetes. Scores range from 8 (not confident at all) to 80 (totally confident).
Diabetes Self-Management Questionnaire scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in ability to self manage diabetes- related activities. The Diabetes Self-Management Questionnaire will be used to assess effective self-care behaviour, with a score of 0 indicating least effective self-care behaviour and 10 indicating most effective self-care.
Problem Areas in Diabetes Scale scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in Diabetes Scale scores. The Problem Areas in Diabetes Scale will assess emotional distress related to diabetes. Scores can range from 0-100, with scores above 40 indicating higher levels of emotional burnout and scores below 10 indicating denial when combined with poor glycemic control.
EQ-5D-5L scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in self-reported overall health. The EQ-5D-5L is a 5-item tool that will be used to assess health factors such as mobility, self care, usual activities, pain, anxiety. Level 1 scores indicate "no problems", levels 2-4 scores indicate more frequent problems, level 5 indicates extreme impairments.
Hypoglycemic Episodes | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in frequency of hypoglycemic episodes. Frequency of hypoglycemic episodes is measured using a single question ("In the past year, how many times have you had a severe low blood sugar reaction, such as passing out or needing help to treat the reaction?"). Categorical responses include 0, 1-3, 4-6, 7-11, 12 or more. Severe hypoglycemia is indicated at 4 or more times.
Barriers to Care for People with Chronic Health Conditions scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in barriers to care. The Barriers to Care for People with Chronic Health Conditions - Economic Barriers to Care scale and Insurance scale will assess economic related barriers in accessing care, which includes services, equipment, and/or medication. Responses of "always", "often", or "sometimes" indicate economic barriers are present.
Health Canada's Household Food Security Survey Module scores | Assessed at Baseline (0 months) and Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in experiences of household food insecurity. Health Canada's 18-item Household Food Security Survey Module will be used to assess experiences of marginal (1 affirmative response), moderate (2-5 affirmative responses) and severe (≥ 6 affirmative responses) household food insecurity in the past 6 months.
Diabetes Competing Demands scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in Diabetes Competing Demands scores. The Diabetes Competing Demands 2-item scale will be used to assess the frequency of trade-offs between food, medicine, and diabetes supplies. A response of "often" or "sometimes" to either question indicates trade-offs have occurred.

OTHER OUTCOMES:
MacArthur Scale of Subjective Social Status scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in subjective social status. The MacArthur Scale of Subjective Social Status national and community ladders consist of a self-reported visual analog scale, whereby respondents place themselves on a ladder rung according to their perceived social standing relative to others in their nation or community. Responses can take a value from 1-10, with a higher score indicating higher subjective social status in relation to others' within ones' nation or community.
Work Productivity and Activity Impairment scores | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in Work Productivity and Activity Impairment scores. The Work Productivity and Activity Impairment 6-item scale will be used to assess impairments in paid and unpaid work due to health issue(s) in the last 7 days. Four scores are calculated including absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism + presenteeism), and activity impairment. Higher scores in each category indicate greater impairment and less productivity.
Perceived Income Adequacy | Assessed at Baseline (0 months) and Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in perceived income adequacy, which is measured using a single question ("To what extent do you think your income is enough for you to live on?"). Using a 5-point response scale, scores are calculated for each participant to indicate either adequate or inadequate income.
Medication Adherence | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in medication adherence. The Simple 1-item Visual Analog Scale consists of a continuum along which participants indicate how often they have taken their prescribed medication in the last 7 days. Responses range from 0% (none at all), 50% (half of prescribed doses), and 100% (all doses of prescribed medications) with higher values indicating greater medication adherence.
Physical Activity Adherence | Assessed at Baseline (0 months) and Follow-up (12 months)
  Difference between intervention and comparison groups in physical activity adherence. Patients will report on how many days during the past week they did a total of 30 minutes or more of physical activity that was enough to raise their heart rate.
Subgroup analyses | Assessed at Baseline (0 months) and Follow-up (6 months, 12 months, 18 months)
  We will conduct subgroup analyses by gender, severity of food insecurity, rural residence, Indigenous status, baseline A1C (6.5-8.5%, 8.6-12%) and insulin use.
Proportion of energy from ultra-processed foods | Assessed twice at Baseline (0 months) and twice at Follow-up (6 months, 12 months, 18 months)
  Difference between intervention and comparison groups in mean proportion of energy from ultra-processed foods

CONTACTS AND LOCATIONS:
Overall Officials: Dana Olstad, PhD, Principal Investigator — University of Calgary
Locations (1):
- Primary Care Clinics, Multiple Locations, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olstad DL, Beall R, Spackman E, Dunn S, Lipscombe LL, Williams K, Oster R, Scott S, Zimmermann GL, McBrien KA, Steer KJD, Chan CB, Tyminski S, Berkowitz S, Edwards AL, Saunders-Smith T, Tariq S, Popeski N, White L, Williamson T, L'Abbe M, Raine KD, Nejatinamini S, Naser A, Basualdo-Hammond C, Norris C, O'Connell P, Seidel J, Lewanczuk R, Cabaj J, Campbell DJT. Healthy food prescription incentive programme for adults with type 2 diabetes who are experiencing food insecurity: protocol for a randomised controlled trial, modelling and implementation studies. BMJ Open. 2022 Feb 15;12(2):e050006. doi: 10.1136/bmjopen-2021-050006. PMID 35168964

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04725630/SAP_001.pdf